CLINICAL TRIAL: NCT02551315
Title: Microarchitecture, Bone Strength and Fracture Risk in Type 2 Diabetes: the DiabOS Study
Brief Title: Microarchitecture, Bone Strength and Fracture Risk in Type 2 Diabetes
Acronym: DiabOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Christian Meier, Prof. Dr. med., University Hospital, Basel, Switzerland
Other Study IDs: EKNZ 2015-117
Record Dates: First submitted 2015-08-25; First posted 2015-09-16 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes Mellitus; Bone Fractures
Keywords: Intra-cortical pore volume; HR-pQCT; DXA; bone mineral density; bone turnover markers; urinary pentosidine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone trunover markers, parameters re calcium metabolism, HbA1c, Insulin, pentosidine, markers of inflammation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Type 2 diabetics, no fractures: Postmenopausal women and men with T2DM, without prevalent fragility fractures (longitudinal follow-up)
- Type 2 diabetics, prevalent fractures: Postmenopausal women and men with T2DM, with prevalent fragility fractures
- Controls, no fractures: Age and sex-matched non-diabetic controls, without fragility fractures (longitudinal follow-up)
- Controls, prevalent fractures: Age and sex-matched non-diabetic controls

SUMMARY:
This multicenter, prospective, observational cohort study will assess bone differences in women and men with type 2 diabetes mellitus (T2DM) with and without fragility fractures.

DETAILED DESCRIPTION:
Cross-sectional evaluation of clinical, biochemical and microstructural measures of bone in patients with type 2 diabetes and age-matched healthy controls. Longitudinal assessment of clinical, biochemical and microstructural measures of bone in study participants without prevalent fragility fractures.

ELIGIBILITY:
Inclusion Criteria:

- presence of type 2 diabetes for at least 3 years (history of treatment for type 2 diabetes)

Exclusion Criteria:

* immobility
* coexisting metabolic bone disease or comorbidities affecting bone health
* previous treatment with osteoporosis medication or intake of medications known to affect bone metabolism (e.g. steroids) within 6 months prior to enrolment
* thiazolidinedione use

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male diabetics (aged between 50 and 75 years; BMI between 18 and 37 kg/m2) Age- and sex-matched non-diabetic controls
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2016-06; Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Intra-cortical pore volume | 2 years
  Intracortical pore volume using HR-QCT femoral shaft and mid-tibia and HR-pQCT at the distal radius (mm3)

SECONDARY OUTCOMES:
Areal Bone Mineral Density (aBMD) | 2 years
  Areal BMD of the spine, the proximal femur and the distal radius (assessed by DXA)
bone turnover markers | 2 years
  alcaline phosphatase, crosslinks
advanced glycation end products (AGE) | 2 years
  urinary pentosidine levels
Occurence of fractures during follow up | 2 years
  incident fracture history
Volumetric Bone Mineral Densitiy (vBMD) | 2 years
  vBMD of the proximal femur, including trabecular and cortical bone in the femoral neck and Trochanter (assessed by HR-QCT)
Cortical thickness and porosity | 2 years
  assessed by HR-QCT at the caudal Region of the femoral neck or the proximal third of the femoral shaft

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meier, Prof. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (5):
- Switzerland (5):
  - Department of Internal Medicine, Kantonsspital Bruderholz, Binningen, Basel-Landschaft
  - University Department of Internal Medicine, University Basel, Kantonsspital, Aarau, Canton of Aargau
  - Department of Internal Medicine, Kantonsspital Luzern, Lucerne, Canton of Lucerne
  - Department of Medicine, St. Anna Hospital Hirslanden, Lucerne, Canton of Lucerne
  - Division of Endocrinology, Diabetology and Metabolism, University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sewing L, Potasso L, Baumann S, Schenk D, Gazozcu F, Lippuner K, Kraenzlin M, Zysset P, Meier C. Bone Microarchitecture and Strength in Long-Standing Type 1 Diabetes. J Bone Miner Res. 2022 May;37(5):837-847. doi: 10.1002/jbmr.4517. Epub 2022 Mar 8. PMID 35094426
- [Result] Vavanikunnel J, Sewing L, Triantafyllidou M, Steighardt A, Baumann S, Egger A, Grize L, Felix B, Kraenzlin M, Henzen C, Meier C. Determinants of Low Bone Turnover in Type 2 Diabetes-the Role of PTH. Calcif Tissue Int. 2022 Dec;111(6):587-596. doi: 10.1007/s00223-022-01022-7. Epub 2022 Oct 3. PMID 36190530
- [Derived] Baumann S, Sewing L, Traechslin C, Verhagen-Kamerbeek W, Grize L, Kraenzlin M, Meier C. Serum Pentosidine in Relation to Obesity in Patients with Type 2 Diabetes and Healthy Controls. Calcif Tissue Int. 2025 Jan 7;116(1):25. doi: 10.1007/s00223-024-01338-6. PMID 39777548